CLINICAL TRIAL: NCT03339869
Title: Evaluation of the Use of Therapeutic Drug Monitoring in the Management of Infections in Intensive Care Unit Patients.
Brief Title: Therapeutic Drug Monitoring of Anti-infectious Drugs in Intensive Care Unit
Acronym: STP-ATB-REA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-05
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: patient hospitalized in intensive care unit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood sample group (Experimental): Adult patient hospitalized in intensive care unit and treated for infection.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — The blood samples will be taken from the patient's bed and then sent to the clinical pharmacology laboratory of Prof. Blin (DRC, Bat F, Timone Hospital).

SUMMARY:
This research targets four anti-infectives commonly prescribed in intensive care: ceftazidime, cefepime, cefotaxime and meropenem, used for severe infections For patient hospitalized in intensive care unit , there is little or no pharmacokinetic data for these four molecules.

DETAILED DESCRIPTION:
Antibiotics, and especially beta-lactams, are among the most used drugs in the world. The good use of antibiotics and the prevention of selection of resistant strains has been a public health priority for many years. In this context, it is essential to obtain effective antibiotic concentrations at the site of infection. In order to obtain effective concentrations, ceftazidime, cefepime, cefotaxime, piperacillin and meropenem are administered in this population by continuous infusion at high dose. Although beta-lactams are mostly well tolerated, they can cause adverse effects such as severe neurological toxicities.

The critically ill patient has physiological alterations that can significantly alter the pharmacokinetics of drugs. Several studies have clearly shown that the pharmacokinetics of beta-lactams in the critically ill patient is different from those of other patients. Depending on the clinical context and the co-morbidities of the patient, sub-therapeutic or potentially toxic concentrations can be observed for the same dosage. The risk of ineffective treatment and the development of resistance remains, despite the high doses administered. In addition, this pharmacokinetic variability may be responsible for the observation of toxic concentrations and the occurrence of adverse effects in this population.

Following these arguments, therapeutic drug monitoring (TDM) of beta-lactams accompanied by personalized dosage adjustment appears to be an essential tool to optimize the management of critically ill patients. Although strongly recommended, the TDM of beta-lactams in the critically ill patient accompanied by a dosage adjustment is not currently performed systematically in all patients.

The objective of this study is to evaluate the impact of the use of a systematic therapeutic drug monitoring of beta-lactams in the critically ill treated with cefotaxime, ceftazidime, cefepime, meropenem or piperacillin, in terms of efficacy and prevention of neurotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age> 18 years)
* Patient hospitalized in intensive care for a duration greater than 7 days, treated with cefotaxime, ceftazidime, cefepime, piperacillin or meropenem according to a standardized dosing regimen.

Exclusion Criteria:

* Age <18
* Pregnant woman
* Patient allergic to beta-lactams
* No written informed consent by the patient or his/her (legal) representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-01-02 (Estimated); Primary Completion 2020-06-02 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
dosage of betalactamins concentrations | 14 days
  Target concentrations are determined from the PK/PD target defined for betalactamins in the intensive care patient, ie a steady-state concentration 100% of the time at 4-5xMIC.

SECONDARY OUTCOMES:
efficacy of the treatment with the clinical response at the end of treatment | 14 days
  Evaluate the efficacy of the treatment with the clinical response at the end of treatment and/or J14 according to the criteria of "resolution / improvement / failure" according to De Waele et al. (Intensive Care Medicine 2014 Sep; 40 (9): 1340-51)

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille

REFERENCES:
- [Derived] Zalta A, Trebuchon A, Daquin G, Velly L, Leone M, Blin O, Lagarde S, Guilhaumou R. Neural correlates of beta-lactam exposure in intensive care unit patients: an observational, prospective cohort study. J Neurol. 2025 Apr 7;272(5):320. doi: 10.1007/s00415-025-13067-3. PMID 40192838